CLINICAL TRIAL: NCT04427878
Title: Is Adipose Tissue a Reservoir for SARS-Cov2 Spread?
Brief Title: Is Adipose Tissue a Reservoir for SARS-Cov2 Spread in Covid-19 Patients?
Acronym: TA/SARS-Cov2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-PP-15
Record Dates: First submitted 2020-06-10; First posted 2020-06-11 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2023-11

CONDITIONS: Covid-19 Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with Covid-19 (Experimental)
  Interventions: Procedure: biopsies of subcutaneous adipose tissue

INTERVENTIONS:
Procedure: biopsies of subcutaneous adipose tissue — Two 4mm punch biopsies of subcutaneous abdominal or thight adipose tissue

SUMMARY:
Resident cells of human adipose tissue express ACE2 and DPP4, receptors for SARS-Cov2. The hypothesis is that the virus may enter and spread in fat depots.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years old
* Patients testing positive for Covid19
* Patients affiliated to social security
* Signing of free and informed consent

Exclusion Criteria:

* Vulnerable persons (- minors,
* adults under guardianship or curatorship,
* pregnant women,
* persons deprived of their liberty,
* persons who do not master the French language)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
The presence of SARS-CoV2 in adipose tissue of Covid19 patients | Day 0
  RT-qPCR for SARS-Cov-2 from RNAs and by immunodetection

SECONDARY OUTCOMES:
The expression of inflammatory cytokines in adipose tissue of Covid19 patients | Day 0
  RT-qPCR for IL6
The expression of inflammatory cytokines in adipose tissue of Covid19 patients | Day 0
  RT-qPCR for IL1
The expression of inflammatory cytokines in adipose tissue of Covid19 patients | Day 0
  RT-qPCR for TNFa

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France